CLINICAL TRIAL: NCT00828490
Title: Developing a Utah Pharmacotherapy Risk Management System With an Electronic Surveillance Tool (Utah ePRM)
Brief Title: Electronic Pharmacotherapy Risk Management
Acronym: ePRM
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Utah Department of Health (Other)
Responsible Party: Jonathan Nebeker MD, University of Utah
Other Study IDs: 24987; 7570516-1
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Last update posted 2010-03-23 (Estimated); Status verified 2010-03

CONDITIONS: Asthma; Mental Health; Pain
Keywords: Fraud and Abuse; opioids
MeSH Terms: conditions — Asthma; Psychological Well-Being; Pain

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Pediatric Asthmatics: Medicaid beneficiaries ≤21 years of age who meet the HEDIS criteria for persistent asthma
  Interventions: Behavioral: provider feedback; Behavioral: patient intervention; Behavioral: Process-level
- Antipsychotic Therapy: Medicaid beneficiaries ≥18 years of age and enrolled ≥6 months of the past 12 months with enrollment in at least one of the past 3 months and ≥3 antipsychotic Rx within past 12 months
  Interventions: Behavioral: provider feedback; Behavioral: patient intervention; Behavioral: Process-level
- Bipolar Therapy: Medicaid beneficiaries ≥18 years of age and enrolled ≥6 months of the past 12 months with enrollment in at least one of the past 3 months and a diagnosis of Bipolar in past 3 years, and ≥ 1 antidepressant Rx in past 6 months, and no mood stabilizer in past 6 months.
  Interventions: Behavioral: provider feedback; Behavioral: patient intervention; Behavioral: Process-level
- Opioid Therapy: Medicaid beneficiaries ≥18 years and enrolled ≥6 of prior 12 months with enrollment in ≥1 of prior 3 months and ≥1 opioid fill in prior 3 months and none of the following in prior 12 months:
  Hospice CPT code or Primary diagnosis of cancer or Oncology CPT code
  Interventions: Behavioral: Process-level
- Fraud and Abuse: Medicaid beneficiaries who filled at least 3 opioid Rx in the last 12 months
- Pediatric Antipsychtotic Therapy: Medicaid beneficiaries <18 years of age with at least 3 antipsychotic Rx's in the past year.

INTERVENTIONS:
Behavioral: provider feedback — The provider-level intervention includes a targeted review of trigger-flagged beneficiaries' drug utilization history and an information packet sent to providers which includes patient-specific pharmacy and medical claims history, patient specific recommendations, and provider comparative profiling.
  Groups: Antipsychotic Therapy; Bipolar Therapy; Pediatric Asthmatics
Behavioral: patient intervention — The patient intervention arm includes the provider-level intervention mentioned above in addition to Medication Therapy Management Services (MTMS), a program that provides patients one-on-one therapy counseling administered by community pharmacists who have completed an MTMS certificate program.
  Groups: Antipsychotic Therapy; Bipolar Therapy; Pediatric Asthmatics
Behavioral: Process-level — The process-level intervention includes the provider-level intervention plus in-clinic evidence-based quality improvement workshops with opportunity for CME credit
  Groups: Antipsychotic Therapy; Bipolar Therapy; Opioid Therapy; Pediatric Asthmatics

SUMMARY:
The purpose of the Utah ePRM (electronic Pharmacotherapy Risk Management) project is to improve quality and safety of medication use while simultaneously controlling costs and detecting fraud and abuse.

DETAILED DESCRIPTION:
The ePRM project has two objectives:

1. Refine and implement a computerized surveillance and trigger tool to support medication therapy and risk management services. The ePRM tool will be used to (1) identify potential drug-therapy problems, which include quality, safety and cost-related problems; (2) select patients and providers for in-depth clinical reviews and possibly direct intervention (i.e., letter, phone call, Medication Therapy Management Services (MTMS), or Academic Detailing); (3) identify potential fraud and diversion of controlled substances; and (4) track patterns of medication use and evaluate ePRM performance, identify improvements, and direct policy change.
2. Conduct innovative multi-pronged interventions that are guided by the ePRM trigger tool. Clinical areas chosen for review include diabetes therapy, hypertension, asthma, antipsychotic therapy, pain management (opioid narcotics and anticonvulsants) and anticoagulation/antiplatelet drugs. Interventions in these areas will address potential under and overuse, or patient safety concerns. Clinical pharmacists and physicians will implement five types of inter-related interventions: a) provider level reviews, which includes prescribers' profiling and feedback for outlier prescribers; b) patient level reviews and letters to prescribers for high-risk patients; c) phone consultation and Academic Detailing with outlier prescribers; d) MTMS; and e) detecting and pursuing suspected fraud and abuse cases.

ELIGIBILITY:
Inclusion Criteria:

* All medicaid recipients and providers with in the salt lake area

Exclusion Criteria:

* each participant much be a Medicaid recipient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all medicaid recipients in the salt lake area
Sampling Method: Non-Probability Sample
Enrollment: 174000 (Actual)
Dates: Start 2007-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan R Nebeker, M.D., M.S., Principal Investigator — VASLCHCS; Gary Oderda, PharmD, M.P.H., Principal Investigator — University of Utah
Locations (1):
- Multi-clinic site, Salt Lake City, Utah, United States